CLINICAL TRIAL: NCT02699645
Title: Triple Therapy Prevention of Recurrent Intracerebral Disease EveNts Trial (TRIDENT), Substudies: MRI, Cognitive
Brief Title: Triple Therapy Prevention of Recurrent Intracerebral Disease EveNts Trial
Acronym: TRIDENT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: The University of New South Wales (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TRIDENT-1103886
Record Dates: First submitted 2016-03-02; First posted 2016-03-04 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Intracerebral Haemorrhage (ICH); Hypertension
Keywords: Blood Pressure (BP); Stroke
MeSH Terms: conditions — Cerebral Hemorrhage; Hypertension; Stroke | interventions — Telmisartan; Amlodipine; Indapamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Triple Pill (active treatment) (Experimental): telmisartan 20mg, amlodipine 2.5mg, and indapamide 1.25mg;
  Interventions: Drug: telmisartan 20mg, amlodipine 2.5mg, and indapamide 1.25mg
- Placebo (Placebo Comparator): Matched placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: telmisartan 20mg, amlodipine 2.5mg, and indapamide 1.25mg — 1 pill taken orally once daily for average of 72 months
  Other Names: Triple Pill
  Arms: Triple Pill (active treatment)
Drug: Placebo — 1 pill taken orally once daily for average of 72 months
  Arms: Placebo

SUMMARY:
An investigator initiated and conducted, multicentre, international, double-blinded, placebo-controlled, parallel-group, randomised controlled trial to determine the effect of more intensive blood pressure control provided by a fixed low-dose combination blood pressure lowering pill ("Triple Pill") strategy on top of standard of care, on time to first occurrence of recurrent stroke in patients with a history of stroke due to intracerebral haemorrhage.

DETAILED DESCRIPTION:
Intracerebral haemorrhage (ICH) is the most serious and least treatable form of stroke, accounting for at least 10% of the 20 million new strokes that occur globally each year. Survivors of ICH are at high risk of recurrent ICH and other serious cardiovascular events.

While there is strong evidence that this risk can be reduced by lowering the blood pressure (BP) of patients after ICH, many patients with ICH do not receive BP-lowering treatment long-term unless BP levels are particularly high, and many do not receive BP combination therapy.

The aim of this study is to assess the safety and efficacy of a combination of fixed low-dose generic BP lowering agents, as a "Triple Pill" strategy on top of standard of care for the prevention of recurrent stroke in patients with a history of ICH and high normal or low grade hypertension. The study is a large-scale, international, double-blind, placebo-controlled, randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with a history of primary ICH that is confirmed by imaging (copy of the brain imaging report to be uploaded to the database, labelled with participant identification (ID) and with personal identifiers removed)
* Clinically stable, as judged by investigator
* Average of two resting SBP levels measured 5 minutes apart in the range 130-160mmHg recorded in a seated position (National Heart Foundation of Australia Guidelines). (Patients with higher SBP can be included if considered by attending clinician that management is consistent with local standards of clinical practice)
* Geographical proximity to the recruiting hospital and/or follow-up medical clinic site to allow ready access for in-person clinic visits during follow-up
* No clear contraindication to any of the study treatments
* Provision of written informed consent

Exclusion Criteria:

* Taking an ACE-I that cannot be switched to any of the following alternatives:

  * telmisartan 20 or 40mg, amlodipine 2.5 or 5mg, indapamide 1.25mg, or
  * an equivalent class (ARB, CCB or thiazide [TZ]-like diuretic), or
  * a BB
* Contraindication to any of the study medications, in the context of currently prescribed BP-lowering medication
* Unable to complete the study procedures and/or follow-up
* Females of child-bearing age and capability, who are pregnant or breast-feeding, or those of child-bearing age and capability who are not using adequate birth control
* Significant hyperkalaemia and/or hyponatremia, in the opinion of the responsible physician
* Estimated glomerular filtration rate (eGFR) <30mL/min/1.73m2
* Severe hepatic impairment (alanine aminotransferase [ALT] or aspartate aminotransferase [AST] >3x the upper limit of normal [ULN])
* Any other condition that in the opinion of the responsible physician or investigator renders the patient unsuitable for the study (e.g. severe disability [i.e. simplified modified Rankin Scale (smRS) of 4-5] or significant memory or behavioural disorder)

Exclusion Criteria for MRI (as applies)

• Any MRI contraindication (e.g. metallic implants, claustrophobia, etc) or participant refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1671 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
Recurrent Stroke | Average of 6 years
  Time to first occurrence of recurrent stroke, whether ischaemic or haemorrhagic.

SECONDARY OUTCOMES:
Recurrent ICH | Average of 6 years
  Time to first occurrence of recurrent ICH
Ischaemic Stroke | Average of 6 years
  Time to first occurrence of ischaemic stroke
Fatal or disabling stroke | Average of 6 years
  Time to first occurrence of fatal or disabling stroke
Mortality | Average of 6 years
  Mortality
MACE | Average of 6 years
  Major adverse cardiovascular events - CV death, non-fatal MI or non-fatal stroke
Physical function | Average of 6 years
  Physical function as assessed by smRS
Change in SBP | Average of 6 years
  Change in SBP
HRQoL according to the EQ-5D-3L | Average of 6 years
  Health-related quality of life according to the European Quality of Life 5-Dimensional Assessment, 3-Level version
Cognitive Impairment | Average of 6 years
  Overall defined by standard cut-points on the Montreal Cognitive Assessment (MoCA)
Cognitive Impairment Supplement | Average of 6 years
  Overall defined by standard cut-points with Brief Memory and Executive Test (BMET) together with assessments of functional impairment related to cognition defined by QDRS score and short form IQCODE, which will also allow subtyping of 'probable' or 'definite' dementia or mild cognitive impairment according to standard diagnostic criteria.
Depression | Average of 6 years
  According to standard cut-point scores on the PHQ-9
Cerebral small vessel disease | Average of 6 years
  Defined by various standard markers on routine MRI, measured by individual components and overall CSVD burden. The primary measure of CSVD is FLAIR WMH volume.
Medication Adherence | Average of 6 years
  Self-reported measures, pill counts
Safety in terms of Serious Adverse Events (SAEs) | Average of 6 years
  SAEs
Tolerability in terms of Adverse Events of Special Interest (AESIs) | Average of 6 years
  AESIs: Headache, Syncope/collapse, Falls, Pedal oedema/ankle swelling, Hypo/hyperkalaemia, Hyponatraemia

CONTACTS AND LOCATIONS:
Overall Officials: Craig Anderson, Principal Investigator — The George Institute
Locations (58):
- Australia (7):
  - Liverpool Hospital, Liverpool, New South Wales
  - Port Macquarie Base Hospital, Port Macquarie, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Brazil (10):
  - Hospital das Clínicas de Botucatu, Botucatu
  - Instituto Flumignano de Medicina, Curitiba
  - Hospital Geral de Fortaleza, Fortaleza
  - Clínica Neurológica e Neurocirurgica de Joinville, Joinville
  - Hospital das Clínicas de Porto Alegre, Porto Alegre
  - Hospital Moinhos de Vento, Porto Alegre
  - Hospital das Clínicas de Ribeirão Preto, Ribeirão Preto
  - Hospital de Base São José do Rio Preto, Rio Prêto
  - Hospital da Bahia, Salvador
  - Universidade Federal de São Paulo, São Paulo
- Georgia (4):
  - LTD Pineo Medical Ecosystem, Tbilisi
  - The First University Clinic of Tbilisi State Medical University, Tbilisi
  - LTD Urgent Neurological Clinic "Neurology", Tbilisi
  - LTD S. Khechinashvili University Hospital, Tbilisi
- Malaysia (5):
  - University Kebangsaan Malaysia Medical Centre, Hulu Langat
  - Hospital Queen Elizabeth, Kota Kinabalu
  - Hospital Universiti Sains Malaysia, Kubang Kerian
  - Sarawak General Hospital, Kuching
  - Hospital Seberang Jaya, Pulau Pinang
- Netherlands (3):
  - Zuyderland Medical Centre, Heerlen
  - Maastricht University Medical Center, Maastricht
  - Radboud University Medical Center, Nijmegen
- Nigeria (5):
  - University College Hospital Ibadan, Ibadan
  - University of Ilorin, Ilorin
  - Jos University Teaching Hospital, Jos
  - Lagos University Teaching Hospital, Lagos, Lagos
  - Ahmadu Bello University Teaching Hospital, Zaria
- National University Hospital, Singapore, Singapore
- Sri Lanka (11):
  - Kandy Teaching Hospital, Kandy, Kandy
  - Ragama Teaching Hospital, Ragama, Ragama
  - Colombo North Teaching Hospital, Colombo
  - Kalubowila (Colombo South) Teaching Hospital, Colombo
  - National Hospital of Sri Lanka, Colombo
  - Karapitiya Teaching Hospital, Galle
  - Gampaha District General Hospital, Gampaha
  - Jaffna Teaching Hospital, Jaffna
  - Teaching Hospital Kurunegala, Kurunegala
  - Sri Jayewardenepura General Hospital, Nugegoda
  - Peradeniya Teaching Hospital, Peradeniya
- Taiwan (3):
  - Chiayi Chang Gung Memorial Hospital, Chiayi City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- United Kingdom (9):
  - Royal Infirmary Edinburgh, Edinburgh
  - Royal Devon & Exeter Hospital, Exeter
  - Queen Elizabeth University Hospital, Glasgow
  - Victoria Hospital, Kirkcaldy
  - Nottingham City Hospital, Nottingham
  - Salford Royal Hospital, Salford
  - Royal Hallamshire Hospital, Sheffield
  - Royal Stoke University Hospital, Stoke-on-Trent
  - Morriston Hospital, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 2 years after publication of main results
Access Criteria: Bone fide researchers submit protocol to the Research Office of The George Institute for Global Health

REFERENCES:
- [Derived] Anderson CS, Rodgers A, de Silva HA, Martins SO, Klijn CJ, Senanayake B, Freed R, Billot L, Arima H, Thang NH, Zaidi WAW, Kherkheulidze T, Wahab K, Fisher U, Lee TH, Chen C, Pontes-Neto O, Robinson T, Wang J, Naismith S, Song L, Schreuder FH, Lindley RI, Woodward M, MacMahon S, Salman RA, Chow CK, Chalmers J. Triple Therapy Prevention of Recurrent Intracerebral Disease Events Trial: Rationale, design and progress. Int J Stroke. 2022 Dec;17(10):1156-1162. doi: 10.1177/17474930211068671. Epub 2022 Jan 7. PMID 34994269
- [Derived] Li L, Poon MTC, Samarasekera NE, Perry LA, Moullaali TJ, Rodrigues MA, Loan JJM, Stephen J, Lerpiniere C, Tuna MA, Gutnikov SA, Kuker W, Silver LE, Al-Shahi Salman R, Rothwell PM. Risks of recurrent stroke and all serious vascular events after spontaneous intracerebral haemorrhage: pooled analyses of two population-based studies. Lancet Neurol. 2021 Jun;20(6):437-447. doi: 10.1016/S1474-4422(21)00075-2. PMID 34022170